CLINICAL TRIAL: NCT02171871
Title: Effects Of Passive Smoking On The Respiratory System Mechanics Of Healthy Non-Smokers In Different Body Positions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hellenic Anticancer Society (Other)
Collaborators: National and Kapodistrian University of Athens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: PBCS003
Record Dates: First submitted 2014-06-03; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: PASSIVE SMOKING ,; RESPIRATORY SYSTEM MECHANICS,
Keywords: EFFECTS,; PASSIVE SMOKING ,; RESPIRATORY SYSTEM MECHANICS,; DIFFERENT BODY POSITIONS.

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CONTROL GROUP (Experimental): Healthy non-smoking volunteers (18-40 years old) will be subject, after giving their brief medical history, to IOS and to the nitrogen washout test. The IOS will be conducted in four positions (standing, sitting, right and left lateral decubitus), whereas the nitrogen washout test in two (sitting and decubitus).
  Then the subjects will be exposed to a smoking environment for 20 minutes.
  Interventions: Other: exposed to a smoking environment

INTERVENTIONS:
Other: exposed to a smoking environment — Then the subjects will be exposed to a smoking environment for 20 minutes, under a continuous measurement of emitted particles using the SIDEPAK AM510 in Pm level 2,5=250, in a closed space of 20 m3. The passive smoking environment will be achieved via a smoking machine. Afterwards, the subject will again undergo IOS in four positions (standing, sitting, right and left lateral decubitus) and nitrogen washout test in two positions (sitting and decubitus). Thanks to the above mentioned techniques, changes in measured parameters will be evaluated.
  Other Names: EFFECTS OF PASSIVE SMOKING; RESPIRATORY SYSTEM MECHANICS

SUMMARY:
The study will examine changes in the respiratory system mechanics and in respiratory physiology after exposure of subjects to passive smoking. It is about healthy non-smoking volunteers and it will be carried out through the techniques of forced oscillation with Impulse Oscillometry (IOS) technique methodology and nitrogen washout.

The present study will contribute to the understanding of passive smoking consequences on the respiratory system of healthy non-smokers. Thanks to the nitrogen washout technique, changes to closing volume and closing capacity will be examined during measurement in different positions (sitting, decubitus) together with exposure to passive smoking. With IOS methodology, changes in respiratory system resistance in four positions (standing, sitting, right and left lateral decubitus) will be evaluated before and after exposure to a passive smoking environment. Results of the present study are expected to provide interesting information on the changes in measured parameters not only in different positions but also after exposure to smoking.

DETAILED DESCRIPTION:
Methodology

For the current study the following techniques will be used. Impulse Oscillometry (IOS) methodology constitutes a method of studying the respiratory system mechanics, during which the investigators manage to determine the flow resistance, the capacity resistance and the resonant frequency through the application of multifrequent signals. It also offers the possibility of studying the mechanics of central and peripheral respiratory system.

The nitrogen washout technique is a method of indirect measurement of the functional residual capacity, during which exhaled nitrogen is measured after the subject has breathed oxygen of a 100% density. A single breath nitrogen washout contributes to the measurement of closing volume and closing capacity.

Emitted particles, detected in a smoking environment, will be measured with the SIDEPAK AM510, which is a measurement device of particles based on their diameter.

The research will be conducted according to the following procedure. Healthy non-smoking volunteers (18-40 years old) will be subject, after giving their brief medical history, to IOS and to the nitrogen washout test. The IOS will be conducted in four positions (standing, sitting, right and left lateral decubitus), whereas the nitrogen washout test in two (sitting and decubitus).

Then the subject will be exposed to a smoking environment for 20 minutes, under a continuous measurement of emitted particles using the SIDEPAK AM510 in Pm level 2,5=250, in a closed space of 20 m3. The passive smoking environment will be achieved via a smoking machine. Afterwards, the subject will again undergo IOS in four positions (standing, sitting, right and left lateral decubitus) and nitrogen washout test in two positions (sitting and decubitus). Thanks to the above mentioned techniques, changes in measured parameters will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteer, adults, non-smokers

Exclusion Criteria:

* < 18 years old , Current pregnancy, Breastfeeding women.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2013-12 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
change of IOS in four positions (standing, sitting, right and left lateral decubitus) | before exposure (Baseline) and after exposure to passive smoking with a 5 minutes interval at one time point
  IOS methodology constitutes a method of studying the respiratory system mechanics, during which we manage to determine the flow resistance, the capacity resistance and the resonant frequency through the application of multifrequent signals. It also offers the possibility of studying the mechanics of central and peripheral respiratory system.

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis K Behrakis, Professor, Study Chair — Hellenic Anticancer Society
Locations (1):
- Hellenic Anticancer Society, Athens, Attica, Greece

REFERENCES:
- [Background] Behrakis PK, Baydur A, Jaeger MJ, Milic-Emili J. Lung mechanics in sitting and horizontal body positions. Chest. 1983 Apr;83(4):643-6. doi: 10.1378/chest.83.4.643. PMID 6831953
- [Result] Stathopoulou H , Vardavas C, Matsunaga Y , Kairi O , Anagnostopoulos N, Karras P , Agaku I, Loukopoulou A, Tzwrtzi A, Behrakis P. The effect of body position during short term exposure to secondhand smoke on pulmonary resistance and impedance using impulse osscilometry European Conference on Tobacco or Health, Istanbul. March 2014